CLINICAL TRIAL: NCT05767320
Title: Comparison Between Open vs Laparoscopic Repair of Perforated Peptic Ulcer
Brief Title: Open vs Laparoscopic Repair of Perforated Peptic Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Magdy Dawood, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: repair of PPU
Record Dates: First submitted 2022-12-24; First posted 2023-03-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Perforated Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Intervention Model Description: patients presenting with perforated peptic ulcer are divided into two groups ,one group undergoes open exploration and the other group undergoes laparoscopy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open approach for perforated pectic ulcer (Active Comparator): repair of perforated peptic ulcer by open technique (exploration)
  Interventions: Procedure: open repair(exploration)
- lap. approach for perforated peptic ulcer (Active Comparator): repair of perforated peptic ulcer by laparoscopy
  Interventions: Procedure: abdominal laparoscopy

INTERVENTIONS:
Procedure: open repair(exploration) — repair of defect of perforated peptic ulcer and peritoneal decontamination by exploration
  Arms: open approach for perforated pectic ulcer
Procedure: abdominal laparoscopy — repair of defect of perforated peptic ulcer and peritoneal decontamination by laparoscopy
  Arms: lap. approach for perforated peptic ulcer

SUMMARY:
comparison between outcomes of both open and laparoscopic repair of perforated peptic ulcer

DETAILED DESCRIPTION:
With the advent of proton pump inhibitors and Helicobacter pylori (H. pylori) eradication therapy, surgical intervention for peptic ulcer disease (PUD) is limited to perforated ulcers in the emergent setting. Perforation is an acute life threatening complication of PUD and occurs in nearly 20% of cases of duodenal ulcer patients . Perforation is a common complication of PUD, with an average 2-14% of peptic ulcers resulting in perforation .While bleeding is the most frequent complication of PUD, perforation carries a higher rate of surgical intervention and is the most lethal complication, associated with a 30-days mortality risk ranging from 3-40%, with advanced age, higher American Society of Anesthesiologists (ASA) classification , elevated body mass index (BMI), and perforation diameter being non-modifiable risk factors associated with increased mortality .The only modifiable risk factor associated with mortality is time to operation, whereby a delay of more than three hours is associated with a doubling of mortality risk .In the 1990s, laparoscopic repair of PPUs was first described . Laparoscopy allows for minimally invasive detection and closure of the lesion with adequate peritoneal lavage, without the drawbacks of an upper laparotomy .Less postoperative pain and analgesic consumption, shorter recovery durations, and decreased wound infections are just some of the advantages of laparoscopic repair . The choice of surgical technique, laparoscopy versus laparotomy, varies depending on the patient's preoperative clinical status, surgeon expertise/preference, and location of defect, with the goal of short operative time. It has been widely reported that open abdominal surgery increases postoperative pain and is associated with higher morbidity (ventral incisional hernia rate, surgical site infection, postoperative respiratory compromise, delayed recovery times, and dehiscence) when compared to laparoscopic surgery . Laparoscopy allows for minimally invasive detection and closure of the lesion with adequate peritoneal lavage, without the drawbacks of an upper laparotomy. Less postoperative pain and analgesic consumption, shorter recovery durations, and decreased wound infections are just some of the advantages of laparoscopic repair .Despite these favorable outcomes, laparoscopic repair is less commonly used, owning to longer operative times in less experienced centers, higher incidence of reoperations owning to leakage at the repair site, and higher incidence of intraabdominal fluid collections secondary to inadequate lavage and the requirement of extensive surgical skill . Additionally, others point to laparotomy as the better treatment, especially for repairing ulcers larger than 9 mm.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 16 years old and younger than 70 years old.
* Patients presenting with acute abdomen due to perforated peptic ulcer
* Patients eligible for laparoscopic surgeries

Exclusion Criteria:

* Patients younger than 16 years old and older than 70 years old
* Contraindications to laparoscopic surgeries as (Hemodynamic instability/shock, Acute intestinal obstruction with dilated bowel loops, Increased intracranial pressure, Relative contraindications, Cardiac failure, Pulmonary failure, Pregnancy/large pelvic masses, Soft tissue infection at port sites, Expected (extensive) adhesions from a previous abdominal surgery)
* Patients who absconded or left the study or died during the period of study.
* Patients with a surgical diagnosis other than perforated peptic ulcer

Ages: 17 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
short term outcomes of both open and lap. Repair of perforated peptic ulcer; operative time | baseline
  comparison of operative time of both laparoscopic and open surgical repair of perforated peptic ulcer
short term outcomes of both open and lap. Repair of perforated peptic ulcer; repair site leakage | baseline
  comparison of repair site leakage between both lap. and open surgical repair of perforated peptic ulcer by follow up through drains inspection.
short term outcomes of both open and lap. Repair of perforated peptic ulcer; intra-abdominal abscess | baseline
  comparison of intra-abdominal abscess formation between both lap. and open surgical repair of perforated peptic ulcer by follow up through abdominal ultrasonography.
short term outcomes of both open and lap. Repair of perforated peptic ulcer; surgical site infection | baseline
  comparison of surgical site infection between both lap. and open surgical repair of perforated peptic ulcer through daily dressing and wound inspection for signs of inflammation.
short term outcomes of both open and lap. Repair of perforated peptic ulcer; postoperative ileus | baseline
  comparison of postoperative ileus between both lap. and open surgical repair of perforated peptic ulcer by follow up of bowel movements.
short term outcomes of both open and lap. Repair of perforated peptic ulcer; hospital stay | baseline
  comparison of duration of patient's hospital stay between both lap. and open surgical repair of perforated peptic ulcer.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Mohamed, Mch, Study Chair — Assiut university hospitals; Mostafa Sayed, Mch, Study Director — Assiut university hospitals; Ibrahim Mostafa, Mch, Study Director — Assiut university hospitals
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Bertleff MJ, Lange JF. Laparoscopic correction of perforated peptic ulcer: first choice? A review of literature. Surg Endosc. 2010 Jun;24(6):1231-9. doi: 10.1007/s00464-009-0765-z. Epub 2009 Dec 24. PMID 20033725
- [Background] Chung KT, Shelat VG. Perforated peptic ulcer - an update. World J Gastrointest Surg. 2017 Jan 27;9(1):1-12. doi: 10.4240/wjgs.v9.i1.1. PMID 28138363
- [Background] Wang YR, Richter JE, Dempsey DT. Trends and outcomes of hospitalizations for peptic ulcer disease in the United States, 1993 to 2006. Ann Surg. 2010 Jan;251(1):51-8. doi: 10.1097/SLA.0b013e3181b975b8. PMID 20009753
- [Background] Soreide K, Thorsen K, Harrison EM, Bingener J, Moller MH, Ohene-Yeboah M, Soreide JA. Perforated peptic ulcer. Lancet. 2015 Sep 26;386(10000):1288-1298. doi: 10.1016/S0140-6736(15)00276-7. PMID 26460663
- [Background] Moller MH, Adamsen S, Thomsen RW, Moller AM; Peptic Ulcer Perforation (PULP) trial group. Multicentre trial of a perioperative protocol to reduce mortality in patients with peptic ulcer perforation. Br J Surg. 2011 Jun;98(6):802-10. doi: 10.1002/bjs.7429. Epub 2011 Mar 25. PMID 21442610
- [Background] Svanes C, Lie RT, Svanes K, Lie SA, Soreide O. Adverse effects of delayed treatment for perforated peptic ulcer. Ann Surg. 1994 Aug;220(2):168-75. doi: 10.1097/00000658-199408000-00008. PMID 8053739
- [Background] Mouret P, Francois Y, Vignal J, Barth X, Lombard-Platet R. Laparoscopic treatment of perforated peptic ulcer. Br J Surg. 1990 Sep;77(9):1006. doi: 10.1002/bjs.1800770916. No abstract available. PMID 2145052
- [Background] Arnaud JP, Tuech JJ, Bergamaschi R, Pessaux P, Regenet N. Laparoscopic suture closure of perforated duodenal peptic ulcer. Surg Laparosc Endosc Percutan Tech. 2002 Jun;12(3):145-7. doi: 10.1097/00129689-200206000-00001. PMID 12080252
- [Background] Lau H. Laparoscopic repair of perforated peptic ulcer: a meta-analysis. Surg Endosc. 2004 Jul;18(7):1013-21. doi: 10.1007/s00464-003-8266-y. Epub 2004 May 12. PMID 15136924
- [Background] Bertleff MJ, Halm JA, Bemelman WA, van der Ham AC, van der Harst E, Oei HI, Smulders JF, Steyerberg EW, Lange JF. Randomized clinical trial of laparoscopic versus open repair of the perforated peptic ulcer: the LAMA Trial. World J Surg. 2009 Jul;33(7):1368-73. doi: 10.1007/s00268-009-0054-y. PMID 19430829
- [Background] Di Saverio S, Bassi M, Smerieri N, Masetti M, Ferrara F, Fabbri C, Ansaloni L, Ghersi S, Serenari M, Coccolini F, Naidoo N, Sartelli M, Tugnoli G, Catena F, Cennamo V, Jovine E. Diagnosis and treatment of perforated or bleeding peptic ulcers: 2013 WSES position paper. World J Emerg Surg. 2014 Aug 3;9:45. doi: 10.1186/1749-7922-9-45. eCollection 2014. No abstract available. PMID 25114715